CLINICAL TRIAL: NCT02044523
Title: Comparison of Magnetic Resonance and Ultrasound Elastography With Liver Biopsy for Noninvasive Staging of Liver Fibrosis
Brief Title: Noninvasive Staging of Liver Fibrosis: MR vs Ultrasound
Acronym: ELF
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: CE12.062
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C; Hepatitis B; Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH)
Keywords: Chronic liver disease; Fibrosis; Elastography; Ultrasound; Magnetic resonance elastography; Diagnostic performance; Sensitivity and specificity
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Non-alcoholic Fatty Liver Disease; Fibrosis; Hypersensitivity | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Liver biopsy specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatis C, Hepatitis B, NAFLD: All patients enrolled will undergo:
  * Transient Elastography (Fibroscan)
  * Acoustic Radiation Force Impulse (ARFI)
  * Magnetic Resonance Elastography (MRE)
  Interventions: Device: Transient elastography, acoustic radiation force impulse, magnetic resonance elastography

INTERVENTIONS:
Device: Transient elastography, acoustic radiation force impulse, magnetic resonance elastography — Transient elastography (Fibroscan) Acoustic Radiation Force Impulse (ARFI) Magnetic Resonance Elastography (MRE)
  Other Names: Transient elastography (Fibroscan); Acoustic Radiation Force Impulse (ARFI); Magnetic Resonance Elastography (MRE)

SUMMARY:
Liver fibrosis is an important public health problem, with a substantial morbidity and mortality due to progression to cirrhosis and hepatocellular carcinoma. All causes of chronic liver disease may lead to fibrosis. The traditional diagnostic approach requires a biopsy for assessing the severity of liver disease prior to therapy.

However, liver biopsy has several limitations: cost, sampling error, and procedure-related morbidity and mortality. Considering the high prevalence of viral hepatitis and nonalcoholic fatty liver disease, a condition often associated with obesity and type 2 diabetes, there is an urgent need for noninvasive screening, diagnosis and monitoring strategies of chronic liver disease severity.

Our team has the expertise to investigate ultrasound-based and magnetic resonance-based elastographic methods for the noninvasive staging of liver fibrosis.

The primary objective of this cross-sectional study is to compare the sensitivity of elastographic methods for detecting histology-determined significant fibrosis.

The secondary objectives are to compare the diagnostic accuracy of these elastographic methods and the influence of potential confounders (inflammation, steatosis and iron deposition) on their diagnostic accuracy.

DETAILED DESCRIPTION:
Background: Liver fibrosis is an important public health problem, with a substantial morbidity and mortality due to cirrhosis (the end stage) and hepatocellular carcinoma. All causes of chronic liver disease may lead to fibrosis. The amount of fibrosis determines the prognosis and influences the response to treatment of chronic liver disease.

Several elastographic methods have been proposed for noninvasive detection and staging of liver fibrosis. Transient elastography (Fibroscan) is widely used by clinicians. Acoustic radiation force impulse (ARFI) is an elastography technique recently integrated in clinical ultrasound systems that may provide similar diagnostic performance to transient elastography. Magnetic resonance elastography (MRE) is a new method that can be integrated to a liver MRI study, which would allow liver stiffness, steatosis, iron overload and inflammation quantification in chronic liver disease.

Objectives: 1) To compare the sensitivity of MRE and ARFI for detecting histology-determined significant fibrosis (F ≥ 2). Secondary objectives: 2) To compare the diagnostic accuracy of MRE, ARFI and Fibroscan for predicting histology-determined fibrosis stages. 3) To determine the influence of inflammation, steatosis, and iron deposition on the diagnostic accuracy of MRE, ARFI and Fibroscan for predicting fibrosis. 4) To determine thresholds optimizing sensitivity of ARFI and Fibroscan to screen patients and optimizing specificity of MRE to confirm liver fibrosis stage.

Design: This will be a cross-sectional imaging trial comparing feasibility, diagnostic and fibrosis staging accuracy of stiffness measurements by elastographic methods in 108 patients with chronic liver disease, using histopathology as the reference standard. Paired index tests (MRE, ARFI and Fibroscan) will be performed as research procedures in close temporal proximity to the reference test (liver biopsy).

Inclusion criteria: consecutive adult patients with known or suspected chronic liver disease secondary to hepatitis B virus, hepatitis C virus, or nonalcoholic fatty liver disease (NAFLD) undergoing a liver biopsy for clinical indications.

Exclusion criteria: any contraindication to MRI, refusal to participate or provide informed consent, pregnant women, any other cause of chronic liver disease than hepatitis B, hepatitis C or NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* are adults;
* must undergo a liver biopsy as part of their clinical standard of care for suspected or known chronic liver disease caused by HBV, HCV or NASH;
* understand French or English instruction;
* Autoimmune Hepatitis

Exclusion Criteria:

* have any contra-indication to MRI (such as claustrophobia, pacemaker, metallic clips for a neurosurgical procedure);
* are pregnant or trying to become pregnant;
* have a weight or girth preventing them from entering the MR magnet bore;
* are unable to understand or unwilling to provide written informed consent for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adults with any of the three main causes of liver fibrosis: HBV, HCV or NASH. For the purpose of this study, we will recruit patients seen at the hepatology clinic of St-Luc Hospital, a tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Histology-determined fibrosis stage | Within 6 weeks of elastographic methods

SECONDARY OUTCOMES:
Fibroscan-determined liver stiffness | Within 6 weeks of liver biopsy
Acoustic Radiation Force Impulse (ARFI)-determined liver stiffness | Within 6 weeks of liver biopsy
Magnetic Resonance Elastography (MRE)-determined liver stiffness | Within 6 weeks of liver biopsy
Magnetic Resonance Imaging (MRI)-based Proton Density Fat Fraction (PDFF) | Within 6 weeks of liver biopsy
Magnetic Resonance Imaging (MRI) cine-tagging of cardiac-induced motion for staging liver fibrosis | Within 6 weeks of liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: An Tang, MD, MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Lefebvre T, Wartelle-Bladou C, Wong P, Sebastiani G, Giard JM, Castel H, Murphy-Lavallee J, Olivie D, Ilinca A, Sylvestre MP, Gilbert G, Gao ZH, Nguyen BN, Cloutier G, Tang A. Prospective comparison of transient, point shear wave, and magnetic resonance elastography for staging liver fibrosis. Eur Radiol. 2019 Dec;29(12):6477-6488. doi: 10.1007/s00330-019-06331-4. Epub 2019 Jul 5. PMID 31278577